CLINICAL TRIAL: NCT04743180
Title: European All-comers' Multicentric Prospective REGISTRY on LUMINOR© Drug Eluting Balloon in the Superficial Femoral Artery and Popliteal Artery With 5 Years Follow-up.
Acronym: LUMIFOLLOW
Status: Recruiting | Type: Observational
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUMIFOLLOW Registry
Record Dates: First submitted 2021-02-01; First posted 2021-02-08 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Angioplasty; Peripheral Arterial Disease; Drug-eluting Balloon; Femoral Artery; Paclitaxel
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUMINOR© drug eluting balloon
  Interventions: Device: LUMINOR© Paclitaxel eluting balloon

INTERVENTIONS:
Device: LUMINOR© Paclitaxel eluting balloon — Patients will be treated with the Luminor paclitaxel eluting balloon

SUMMARY:
The objective of this all-comers registry is to explore the safety, efficacy, and cost-efficiency of the LUMINOR© DEB in de-novo and restenotic-FP lesions. For de-novo and restenotic lesions, especially for calcified and/or long lesions/occlusions, the use of debulking devices to improve recalibration and drug penetration will be evaluated in a specific sub-group.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Rutherford Clinical Category 2-5
* The subject is legally competent, has been informed of the nature, the scope, and the relevance of the study, voluntarily agrees to participation, is willing to provide 5-year informed consent and has duly signed the informed consent form (ICF)
* Significant (≥ 70%) stenosis or occlusion of a native femoropopliteal artery
* TASC II Class A to D Lesions
* de novo lesion(s), non-stented or stented restenotic lesion(s)
* Proximal margin of target lesion(s) starts at the ostium of the superficial femoral artery, just below the common femoral bifurcation
* Distal margin of target lesion(s) terminates at bifurcation of popliteal artery AND ≥1 cm above the origin of the TP trunk (P3)
* A patent inflow artery free from significant lesion (≥ 50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of iliac or common femoral inflow artery lesions); Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤ 30% without death or major vascular complication
* Successful wire crossing and pre-dilatation (1min min, with under sizing of 1mm compared to ref diameter) of the target lesion; Use of crossing devices allowed if necessary. Use of laser or atherectomy is allowed if necessary, during the index procedure. Bailout stenting is allowed if necessary, after DEB use
* At least one patent native outflow artery to the ankle, free from significant (≥ 50%) stenosis as confirmed by angiography (treatment of outflow disease is NOT permitted during the index procedure)

Exclusion Criteria:

* Women who are pregnant, lactating, or planning on becoming pregnant or men intending to father children
* Patient is contraindicated to use Luminor Drug Eluting Balloon per the current Instructions For Use (IFU)
* Life expectancy of < 1year
* Patient is currently participating in an investigational drug or other device study or previously enrolled in this study
* Inability to take required study medications or allergy to contrast that cannot be adequately managed with pre- and post-procedure medication
* Sudden symptom onset, acute vessel occlusion, or acute or sub-acute angiographically visible thrombus in target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery disease due to occlusive lesions, stenosis of ingraguinal arteries and restenosis after previous angioplasty with/without stent in that sector.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint Efficacy measured by presence of primary patency of the target lesion based on ultrasound images | 12 Months
  Primary Patency is defined as Freedom from Clinically-Driven Target Lesion Revascularization and from Binary Restenosis.
Overall Medical Safety | 36 Months
  Combination assessment of freedom from all-cause peri-procedural (≤30 day) death and freedom at 3 years from the following: index limb amputation (above or below the ankle), and all-cause mortality (with a detailed analysis of cardiovascular (CV) and non-CV deaths). Success is defined as freedom from all specified events; failure is defined as one or more specified events occurrences.

SECONDARY OUTCOMES:
Secondary Endpoint Medical Safety: Major vascular complications | ≤30 days after index procedure
  Major vascular complications will be counted:
  * Haematoma at access site >5 cm
  * False aneurysm
  * AV fistula
  * Retroperitoneal bleeding
  * Peripheral ischemia/nerve injury
  * Any transfusion required will be reported as a vascular complication unless clinical indication clearly other than catheterization complication
  * Vascular surgical repair
Secondary Endpoint Medical Safety: Composite Safety | 1, 6, 12, 36, 48, 60 months after index procedure
  Combination assessment of freedom from all-cause death and freedom from the following: index limb amputation (above or below the ankle = major or minor amputation) and index limb re-intervention. Success is freedom from all specified events; failure is occurrence of one or more specified events.
Secondary Endpoint Medical Safety: All-cause death | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Death by any cause will be counted and stratified between CV and non-CV deaths. Cause of death will be analyzed to search for any specific increase of a death's subtype.
Secondary Endpoint Medical Safety: Major amputation at target limb | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Amputations above the ankle of the target leg will be counted. Optional histologic examination of fixed muscle segments in 10% neutral-buffered formalin could be performed in the Inserm unit 1034, Pessac, France to search for paclitaxel microparticle deposits, fibrinoid necrosis artery wall injury, inflammation, thrombus, hemorrhage, and fibrosis. Adjacent nonfixed samples of similar distal tissues, flash-frozen in liquid nitrogen, and retained at -80°C will be used for bioanalysis of paclitaxel levels by modified liquid chromatography/tandem mass spectroscopy.
Secondary Endpoint Medical Safety: Minor amputation at target limb | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Amputations below the ankle of the target leg will be counted.
Secondary Endpoint Medical Safety: Target Vessel Revascularization (TVR) | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Repeat intervention at the target vessel will be counted.
Secondary Endpoint Medical Safety: Target Limb Reintervention | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Repeat intervention at the target leg will be counted.
Secondary Endpoint Efficacy: Acute Device Success | During index procedure
  Device success is defined as, a per device basis, the achievement of successful delivery and deployment of the study device(s) as intended at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the study system. If a device is inserted into the subject but not used due to user error (e.g. inappropriate balloon length or transit time too long), this device will not be included in the device success assessment.
Secondary Endpoint Efficacy: Technical Success | During index procedure
  Technical Success of the balloon procedure is defined as successful access and deployment of the device and visual estimate of ≤ 30% diameter residual stenosis during the index procedure.
Secondary Endpoint Efficacy: Procedural Success | Up to 30 days
  Attainment of ≤ 30% residual stenosis in the treatment area without major adverse events (defined as occurrence of death, major amputation of the target limb, target vessel or distal revascularization) during the index procedure and through the hospital stay.
Secondary Endpoint Efficacy: Primary Patency | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Primary Patency is defined as Freedom from Clinically-Driven Target Lesion Revascularization and from Binary Restenosis. Binary restenosis is adjudicated by the validated center based on threshold Doppler PSVR ≥ 2.5 (together with waveform analysis & color mosaic appearance) or based on angiographic ≥ 50% diameter stenosis (if angiography is performed although not required per protocol).
Secondary Endpoint Efficacy: Secondary Patency | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Secondary Patency of the target lesion is defined as the absence of binary restenosis as adjudicated by the validated center, independent of whether or not patency is re-established via an endovascular procedure.
Secondary Endpoint Efficacy: Clinically-driven Target Lesion Revascularization (TLR) | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Revascularization of the target lesion with evidence of diameter stenosis >50% determined by duplex ultrasound or angiography and new distal ischemic signs (worsening ABI or worsening Rutherford Category associated with the target limb or due to clinical symptoms).
Secondary Endpoint Efficacy: Target Lesion Revascularization (TLR) | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  A repeat revascularization procedure (percutaneous or surgical) of the original target lesion site.
Secondary Endpoint Efficacy: Change of Rutherford classification from baseline | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  Patients are enrolled with a Rutherford grade of 2-5 for their target leg. The Rutherford scale is an indicator for the severity of Peripheral Vascular Disease: 0 = no symptoms, 6 = functional foot is no longer salvageable (leading to foot amputation).
Secondary Endpoint Efficacy: Change of resting Ankle Brachial Index (ABI) from baseline | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  The ABI values will be recorded and compared to the baseline values. The ABI is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm. A ratio of 0.9-1.3 is in the normal range. Lower ratios indicate bad blood perfusion of the leg.
Secondary Endpoint Efficacy: Change in Walking Impairment Questionnaire from baseline | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  The Walking Impairment Questionnaire values will be recorded and compared to the baseline values.
Secondary Endpoint Efficacy: Change in quality of life from baseline, as measured by EQ-5D | 1, 6, 12, 24, 36, 48, 60 months after index procedure
  The EQ-5D Questionnaire values will be recorded and compared to the baseline values.
Secondary Endpoint Cost-Effectiveness (optional): factoring procedure and hospital admission costs | 1, 6, 12, 24, 36, 48, 60 months after index procedure

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Centre Hospitalier Universitaire Pellegrin, Bordeaux, Nouvelle-Aquitaine
  - Clinique Générale Annecy, Annecy
  - Clinique Rhône Durance, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - Polyclinic Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre Hospitalier Régional Universitaire Morvan de Brest, Brest
  - CHRU Lille, Lille
  - Clinic Mutualiste Porte de L'Orient, Lorient
  - CHU Timone Marseille, Marseille
  - CH Layné, Mont-de-Marsan
  - Hôpital Privé des Franciscaines, Nîmes
  - Fondation Hôpital St Joseph, Paris
  - Clinique Saint Jean, Saint-Jean-de-Védas
  - Clinique Rhéna, Strasbourg

IPD SHARING:
Plan to Share IPD: No